CLINICAL TRIAL: NCT01609036
Title: An Observational Phase IV Non Interventional Study in Patients With Advanced Follicular Lymphoma (III-IV) Evaluating the Safety of Maintenance Therapy With Rituximab After 8 Cycles of Rituximab in Combination With Chemotherapy as Induction Therapy in Previously Untreated Patients in Greece.
Brief Title: An Observational Study of MabThera/Rituxan (Rituximab) in Patients With Follicular Lymphoma
Status: Terminated | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22236
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the safety and efficacy of MabThera/Rituxan (rituximab) in previously untreated patients with follicular lymphoma. Data will be collected for 3 years

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years
* Patients with previously untreated follicular lymphoma (stage III-IV) according to the approved summary of product characteristics (SPC)

Exclusion Criteria:

* Contraindications to MabThera/Rituxan therapy according to the approved SPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage III-IV follicular lymphoma
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 3 years

SECONDARY OUTCOMES:
Progression-free survival | 3 years
Event-free survival | 3 years
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Greece (3):
  - Athens
  - Pátrai
  - Thessaloniki